CLINICAL TRIAL: NCT04382833
Title: EFFECTS OF MASSAGE AND HOT APPLICATION ON LABOR PAIN AND COMFORT
Brief Title: MASSAGE AND HOT APPLICATION ON LABOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Hülya TÜRKMEN, Lecturer (PhD), Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BalıkesirU
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Labor Pain
Keywords: comfort at labor; labor pain; hot application; massage
MeSH Terms: conditions — Labor Pain | interventions — Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HOT APPLICATION GROUP (Experimental): Thermoforming, one of the dry hot application methods, was performed on the sacral (S1-S4) vertebrae region of pregnant women in the hot application group while they were in sitting or left-side-lying position (during 4-5, 6-7, and 8-9 cm cervical dilation). Thermoforming was applied by wrapping it with a towel to protect pregnant women from the direct effect of its hot surface. The mean water temperature used in thermoforming was 50C. The water temperature was measured using a liquid thermometer. When 50°C water was subjected to hot application, the surface temperature reached around 40°C. The hot application was carried out continuously for 20 min.20 The body temperature of the pregnant women was evaluated before the application.
  Interventions: Other: HOT APPLICATION
- MASSAGE GROUP (Experimental): Massage using effleurage and friction techniques was applied to the 4-5 cm right and left lateral parts of the midline on the sacral (S1-S4) vertebrae region of pregnant women in the massage application group while they were in sitting or left-side-lying position (during 4-5, 6-7, and 8-9 cm cervical dilation). The massage application was carried out continuously for only 10 min because it was thought to cause irritation to the area where it was practiced.
  Interventions: Other: MASSAGE
- CONTROL GROUP (No Intervention)

INTERVENTIONS:
Other: HOT APPLICATION — HOT APPLICATION
  Arms: HOT APPLICATION GROUP
Other: MASSAGE
  Arms: MASSAGE GROUP

SUMMARY:
Aim: This study aimed to examine the effects of sacral massage and hot application on labor pain and comfort level perceptions in pregnant women.

Methods: This randomized controlled experimental study included hot application, massage and control groups, each having 30 primiparous pregnant women whose cervix was dilated to 4-5 cm. The intervention groups were given a sacral massage or sacral hot application, whereas the control group was given only standard midwifery care during 4-5, 6-7, and 8-9 cm cervical dilation. The data were collected using the Introductory Information Form, the Childbirth Comfort Questionnaire (CCQ), and the Numerical Rating Scale (NRS).

DETAILED DESCRIPTION:
This randomized controlled experimental study was carried out between June and December 2016 in the delivery room of Public Hospital in Turkey.The sample size was determined using power calculations G*Power 3 with taking into account previous studies in which a effects massage and hot application on labor pain. Estimates of effects were derived from the findings of previous studies. The sample size was calculated at the 5% level of significance and a power of 95% based on previous studies (n = 30 in each group). The study sample consisted of primiparous pregnant women with vaginal delivery expectancy, term pregnancy, single healthy fetus, and active labor stage (4-5 cm dilation). A total of 98 primiparous pregnant women were included in the study, but 8 of them were excluded because of delivery by cesarean section. Thus, three research groups were formed as follows: massage, hot application, and control groups (n =30 in each group). Sacral massage and sacral hot application were applied to the intervention groups, and only standard midwifery care was given to the control group. Randomization was performed when each pregnant woman who was admitted to the hospital during labor and met the inclusion criteria. Randomization was provided with the collection of data on Mondays, Wednesdays, and Fridays of each week during the study period. Sacral massage was applied on Mondays, sacral hot application was performed on Wednesdays, and data of the control group were collected on Fridays. Cervical dilation and effacement, contraction, fetal heartbeat rate, and vital findings were followed in the standard midwifery care. Midwives informed pregnant women about breathing and evacuation techniques. In addition, all pregnant women in labor process received induction application. Each study group was given a descriptive information form, Childbirth Comfort Questionnaire (CCQ), and Numerical Rating Scale (NRS) in the active stage of labor (4-5 cm cervical dilation). Standard midwifery care was given to each group, and intervention groups were interfered three times in total, during 4-5, 6-7, and 8-9 cm cervical dilation. Immediately after each intervention, NRS was administered between contractions. CCQ was also applied between contractions after the last intervention made during 8-9 cm cervical dilation. Pregnant women in the control group filled NRS during 4-5 and 6-7 cm cervical dilation, and CCQ during 8-9 cm cervical dilation. NRS was applied for the last time in all three groups 5 min after the third stage of labor.

Childbirth Comfort Questionnaire-CCQ: This scale was developed by Schuling and Sampselle (2003), and the Turkish validity and reliability study of the scale was carried out by Potur et al (2015). Potur et al. (2015) showed that the sociocultural subscale had item total score correlation coefficient less than 0.30, and the items showing the relief level were extracted from the scale. The CCQ consisted of physical, environmental, and psychospiritual subscales and a specific sense of relief and transcendence. It was a 5-point Likert-type scale with nine items. Each item scored between strongly disagree (1 point) to strongly agree (5 points). It is possible to score from 9 to 45 when all questions on the scale are answered. High score referred to high comfort and vice versa. In the present study, CCQ was applied two times in total, one before the intervention during 4-5 cm cervical dilation and one immediately after the intervention during 8-9 cm cervical dilation.

Numerical Rating Scale (NRS): This scale was used to evaluate pain levels.Subjects were asked to rate the level of their pain using the numbers from 0 (no pain) to 10 (worst imaginable pain) on this scale. In the present study, NRS was applied five times in total, one before the intervention, three times immediately after interventions (during 4-5, 6-7, and 8-9 cm cervical dilations) and one after delivery

ELIGIBILITY:
Inclusion Criteria:

* primiparous pregnant women
* vaginal delivery expectancy
* term pregnancy
* single healthy fetus
* active labor stage (4-5 cm cervikal dilation)

Exclusion Criteria:

* multioarous pregnant women
* preterm labor
* multiple pregnancy
* complicated pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant womens
Enrollment: 90 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
severity of labor pain assessed by Numerical Rating Scale | 4-5 cm, 6-7 cm and 8-9 cm cervical dilation at labor
  Labor pain level, Numerical Rating Scale
comfort level at labor | 4-5 cm and 8-9 cm cervical dilation at labor
  Comfort level, Childbirth Comfort Questionnaire

IPD SHARING:
Plan to Share IPD: No